CLINICAL TRIAL: NCT01053871
Title: Propofol Versus Midazolam With Fentanyl for EGD Endomicroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Li-Yanqing, Department of Gastroenterology, Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2009SDU-QILU-G08
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2009-12

CONDITIONS: Gastritis; Functional Dyspepsia
Keywords: normal
MeSH Terms: conditions — Gastritis | interventions — Propofol; Midazolam; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): sedation using propofol
  Interventions: Drug: propofol
- 2 (Experimental): sedation using midazolam with fentanyl
  Interventions: Drug: midazolam with fentanyl

INTERVENTIONS:
Drug: propofol — conscious sedation using propofol
  Arms: 1
Drug: midazolam with fentanyl — conscious sedation using midazolam with fentanyl
  Arms: 2

SUMMARY:
This trial aims to compare the endomicroscopic image quality and sedation efficacy of propofol or midazolam with fentanyl.

ELIGIBILITY:
Inclusion Criteria:

* outpatients attending endomicroscopy
* able to give written informed consent

Exclusion Criteria:

* GI tract malignancy
* coagulopathy
* acute upper digestive tract bleeding
* pregnancy or breast feeding
* allergy to fluorescein sodium
* impaired renal function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
endomicroscopic image quality | 3 months

SECONDARY OUTCOMES:
sedation efficacy outcomes,patient assessment,physician assessment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China